CLINICAL TRIAL: NCT02828059
Title: Continuous Wound Infiltration for Diminution of Post-surgery Pain After Caesarean Section (Dip-Caesar)
Brief Title: Continuous Wound Infiltration for Diminution of Post-surgery Pain After Caesarean Section
Acronym: dip-Caesar
Status: Withdrawn | Type: Observational
Why Stopped: changed drug approval
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZKSJ0095
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Pain
Keywords: Caesarean section
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropivacaine — Surgical wound Infiltration over 48 hours
  Other Names: ReadyFusor

SUMMARY:
A medical approach that warrants continuous and reliable local administration of non-opioid analgesic drugs might substantially improve post-surgery pain management in CS, while decreasing the necessity of staff-dependent invasive procedures and the probability of untoward effects following systemic drug exposure. ReadyfusOR® is a formulation comprising a Ropivacain-loaded single-use pump which has been approved for regional application of the analgesic drug, also comprising obstetric interventions. There is, however, scarce scientific information on the efficacy and benefit of this anesthetic drug formulation for pain management following CS by means of continuous wound infiltration.

DETAILED DESCRIPTION:
During the past decades the rate of Caesarean sections has increased considerably, with Germany following the global trend. When compared to other surgical interventions, Caesarean section is perceived as very painful. Patient-controlled analgesia (PCA) is associated with significantly higher opioid dosage, as compared to cases where the same medication is administered on patient's request as a bolus by the attending staff. Conceivably, patients using PCA reported less painful sensations. Nonetheless, several patients and physicians express reservations concerning the use of opioids for pain management in lactating mothers. Peripheral application of local anesthetics (e.g. as wound infiltration or peripheral nerve blockade) has been shown in several settings to reduce the demand of systemic drug dosage in pain management. The intended effect, however, lasts only for a couple of hours. Feasibility of subsequent bolus drug applications is hampered by ethical concerns (being an invasive procedure) as well as staff strains and cost effectiveness considerations. Hence, a medical device that warrants continuous and reliable administration of local analgesics might substantially improve pain management in obstetric patients. ReadyfusOR® is a medical device that has been approved for use for such purposes.

This study will record the use of the Ropivacaine formulation ReadyfusOR® under real life conditions in a representative sample. Ropivacaine formulation ReadyfusOR® is established as a standard procedure for diminution of post-surgery pain in the Department of Obstetrics of the Jena University Hospital. The gathered information will be used to augment the knowledge about outcomes and safety of the Ropivacaine formulation ReadyfusOR® using for treatment of patients undergoing Caesarean section. Analgesic efficacy will be monitored at defined intervals over an observation period of 48 h post-surgery using patient's subjective ratings of spontaneous and strain-induced pain perception, as well as the demand of auxiliary dosing of standard analgesic treatment.

At the end of surgery and prior to closure of the abdomen the drug infusion catheter of Readyfusor® is inserted subfascially. An initial priming dose of 10 mL of 2mg/mL ropivacain will be injected through the catheter. After the catheter has been primed with the initial loading dose, the Readyfusor® is activated by the surgeon or nurse in the operating room and connected to the wound catheter. As described in the product information, the wound edges are supplied with Ropivacain over 48 h at a rate of 10 mg/hour (5 mL/hr). During the first 48 h post-surgery patients receive standard pain management with Ibuprofen at doses of 600 mg administered in intervals of 8 hours. If the patients are free of pain Ibuprofen application can be reduced as needed. The synthetic opioid Piritramide is used as pain medication on demand for patients who report mild to severe pain defined as 5 or more points on a 10-point-Numeric Rating Scale (NRS). In either available application option - as PCA or a bolus injection by the attending nurse - the dose of Piritramide is limited to 30 mg over 4 hours and each single application are limited to 3mg every 10 minutes.

Maximal intensity of pain at rest and pain due to mobilization (first standing up) will be assessed at intervals of 12, 24 and 48 h after treatment introduction by means of patient's statements plotted on individual numeric rating scales for each endpoint. The primary endpoint focuses on assessing the perceived spontaneous pain intensity at 24 h post-surgery.

Further characterization of the pain-relieving effect of ReadyfusOR® will be provided by the records on the fractional doses of the auxiliary opioid analgesic Piritramide administered within 12, 24 and 48 h post-surgery. The individual time needed for the recovery of mobility will provide an additional tool for treatment effect evaluation.

Finally, NRS-recorded patient's ratings on subjectively perceived satisfaction with the post-surgical pain management will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergent Caesarean section under spinal or general anesthesia
* Medically indicated necessity of post-surgery analgesia
* Signed informed consent
* Body Mass Index above 20 and below 35

Exclusion Criteria:

* Wound drainage application following surgery
* Epidural catheter following surgery
* Planned concurrent surgical Intervention
* Chronic high-dose opioid use (>20 mg oxycodone equivalent daily) over more than 4 weeks prior to surgery
* History of, suspected or present addiction or abuse of illicit drug(s), prescription medicine(s) or alcohol during the preceding 2 years
* Intolerance or allergy to any of the medications planned for use
* Concurrent painful physical conditions that may require analgesic Treatment
* Current or planned administration of Long-acting Opioids, selective Serotonin reuptake Inhibitors, gabapentin, pregabalin or duloxetine within 30 days preceding and7or following surgery
* Use of systemic glucocorticoids (except for induction of fetal lung maturation) within 1 month prior to enrollment
* Uncontrolled anxiety, schizophrenia or other psychiatric conditions which could interfere with the compliance and subjective assessment of Treatment effects (decision at the discretion of the investigator)
* Inability to operate devices for Patient-controlled analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing delivery by elective or emergent Caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximal perceived pain intensity 24 h after surgery | 24 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale

SECONDARY OUTCOMES:
Perceived pain at rest over 12 h after surgery | 12 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale
Perceived pain at mobilization over 12 h after surgery | 12 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale
Perceived pain at rest over 24 h after surgery | 24 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale
Perceived pain at mobilization over 24 h after surgery | 24 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale
Perceived pain at rest over 48 h after surgery | 48 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale
Perceived pain at mobilization over 48 h after surgery | 48 hours
  Subjectively rated pain perception by a 10-point-numeric rating scale
Opioid demand over 12 h after surgery | 12 hours
  Cumulative dosis of Piritramide administered on demand over 12 hours
Opioid demand over 24 h after surgery | 24 hours
  Cumulative dosis of Piritramide administered on demand over 24 hours
Opioid demand over 48 h after surgery | 48 hours
  Cumulative dosis of Piritramide administered on demand over 48 hours
Satisfaction with pain management 24 h after surgery | 24 hours
  Subjectively rated degree of satisfaction with analgesia by 10-point numeric Rating scale

OTHER OUTCOMES:
Adverse events and adverse drug reactions | 48 hours
  Registration of adverse avents and adverse drug reactions over the duration of Ropivacaine administration

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Schleussner, MD, Study Director — Department of Obstetrics, Jena University Hospital

IPD SHARING:
Plan to Share IPD: No
Dissemination of individual participant data is not planned